CLINICAL TRIAL: NCT06018584
Title: Effect of Low-Level Laser Therapy in Wound Healing and Post-Operative Pain Management of Primary Molar Teeth Ex-traction: A Randomized Clinical Trial
Brief Title: Biostimulation After Tooth Extraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hazal Özer (Other)
Responsible Party: Sponsor-Investigator, Hazal Özer, Assist. Prof., Necmettin Erbakan University
Organization: Necmettin Erbakan University (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017-07
Record Dates: First submitted 2023-08-21; First posted 2023-08-30 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Dental Caries in Children; Wound Heal
MeSH Terms: interventions — Tooth Extraction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (Sham Comparator): No application was made after the tooth extraction procedure in the control group.
  Interventions: Other: Tooth extraction
- Low- Level Laser Group (Doctor Smile Wiser) (Experimental): In the Laser group, the diode laser device Doctor Smile Wiser (Wiser, Doctor Smile, Milan, Italy) (Figue 1) with a wavelength of 980 nm and a power of 0.5 W was used for LLLT. During the procedure, the patient, physician, and assistant staff wore protective glasses (Wiser, Doctor Smile, Milan, Italy). With 300 mW of energy, a 400 m tip held 1 cm away from the extraction socket was applied to the extraction socket for 60 seconds from three points determined from the vestibule, lingual/palatal, and occlusal surfaces.
  Interventions: Other: Tooth extraction

INTERVENTIONS:
Other: Tooth extraction — Tooth extractions were performed by a single physician. Topical anesthesia (Xylo-caine, Astra, Södertalje, Switzerland) was applied to the dried mucosa in the area to be lo-calized with the help of an ear stick for 1 minute. Posterior-superior-alveolar nerve block anesthesia and palatal anesthesia were applied for the upper primary molars; Inferi-or-alveolar nerve block anesthesia and lingual anesthesia (Ultracain, Aventis Pharma, Is-tanbul, Turkey) were applied for the lower primary molars. After anesthesia control was achieved, a randomly selected tooth was extracted. Tooth extraction on the other side was performed two weeks later. During the shootings, attention was paid to the traumatic ap-proach. After the control of bleeding was achieved, data were recorded for each group.

SUMMARY:
This study evaluated the effect of low-level laser therapy on postoperative pain and wound healing in children undergoing primary molar extractions 40children, 6-10 years of age, systemically healthy, and had atraumatic extraction indications of bilateral primary molar teeth were included in the study. A randomly selected tooth was extracted under local anesthesia in the first session. Only the clot formation on the socket was observed and photographed in the control group. Other group extractions were performed 2weeks later. The LLLT group was treated with a 980 nm wavelength Doctor Smile Wiser diode laser and photographed. Non-epithelialized surface measurements were performed with the ImageJ program. Pain assessment was performed with the Wong-Baker Pain Scale. Statistical analyses were performed with SPSS software.

ELIGIBILITY:
Inclusion Criteria:

* indication for tooth extraction in bilateral primary molars
* did not have any systemic disease
* the use of antibiotics and painkillers was stopped at least 12 hours ago

Exclusion Criteria:

* require complicated tooth extractions
* systemic disease
* the use of antibiotics and painkillers in 12 hours

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Wound healing | intervention (tooth extraction) day, 3rd day and 7th day
  For the evaluation of soft tissue healing in extraction sockets, intraoral photographs were taken at an angle of 60° to the occlusal surface on the 3rd and 7th days following the extraction session. Non-epithelialized surface measurements were made by two observing physicians using the ImageJ (NIH, Rockville, USA) program.
Pain score | intervention day (tooth extraction), 3rd day and 7th day
  Pain assessment in both groups was performed with the Wong-Baker Pain Rating Scale (Wong-Baker FACES Pain Rating Scale PRS). Patients were asked to choose a face or number from the scale, and the selected value was the practitioner dentist on the day of the procedure; other days were recorded by the parent. This scale is graded from 0 to 10. 0 indicates no pain, and 10 marks the most severe pain. It is asked to evaluate the pain according to the facial expression.

IPD SHARING:
Plan to Share IPD: Yes
The IPD can be shared when the paper is published.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: From 2024 January for five years
Access Criteria: The e-mail requests will be considered.